CLINICAL TRIAL: NCT05390307
Title: Obesity Treatment to Improve Diabetes
Acronym: OTID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dasman Diabetes Institute (Other)
Responsible Party: Principal Investigator, Dr. Ebaa Al Ozairi, Principal Investigator, Dasman Diabetes Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RA-HM2021009
Record Dates: First submitted 2022-05-14; First posted 2022-05-25 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes Mellitus; Obesity; Chronic Kidney Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Obesity; Renal Insufficiency, Chronic | interventions — Liraglutide; semaglutide; dapagliflozin

STUDY DESIGN:
Intervention Model Description: In this 6-month randomized control trial, 60 participants aged between 21-65 years, with a body mass index (BMI) above 25kg/m2 and T1D with CKD will be randomised to receive one of five possible treatments 1) Standard care (control), 2) GLP1RA alone, 3) SGLT2i alone, 4) combination of GLP1RA and SGLT2i, 5) combination of GLP1RA and SGLT2i with intensive lifestyle advice.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- GLP1RA alone (Experimental): Participants in the GLP1RA will be prescribed either Liraglutide 3.0mg or Semaglutide 1.0mg, whichever is licensed and available locally. The dose and titration will follow the usual clinical practice. The treatment will continue for 6 months.
  Interventions: Drug: Liraglutide / Semaglutide
- SGLT2i alone (Experimental): Participants in the SGLT2i group will be prescribed dapagliflozin 5-10mg once daily for 6 months.
  Interventions: Drug: Dapagliflozin
- GLP1RA/SGLT2i combination (Experimental): Participants in the combination GLP1RA and SGLT2i group will be prescribed liraglutide 3mg once daily or semaglutide1mg once weekly subcutaneous injection plus dapagliflozin 5-10mg for 6 months.
  Interventions: Drug: Liraglutide or Semaglutide / Dapagliflozin
- GLP1RA/SGLT2i combination with intensive lifestyle changes (Experimental): Participants in the combination GLP1RA and SGLT2i and intensive weight loss groupwill be prescribed liraglutide 3mg once daily or semaglutide 1mg once weekly subcutaneous injection plus dapagliflozin 5-10mg together with an intensive dietary and lifestyle approach for 6 months. This typically involves dietary advice to reduce energy intake (and may includea period of partial or total meal replacement), accompanied -if available -by a physical activity programme, both supported by behavioural change techniqueswith regular professional contacts.
  Interventions: Drug: Liraglutide or Semaglutide / Dapagliflozin plus intensive weight loss nutrition
- Usual Care (Experimental): Participants in the usual care arm will follow the best medical care by following the international guidelines for 6 months. This usually involves diet and exercise advice.
  Interventions: Other: Usual care

INTERVENTIONS:
Drug: Liraglutide / Semaglutide — Liraglutide 3mg once daily or semaglutide 1mg once weekly subcutaneous injection for 6 months.
  Other Names: GLP1RA alone
  Arms: GLP1RA alone
Drug: Dapagliflozin — Dapagliflozin 5-10 mg once daily for 6 months.
  Other Names: SGLT2i alone
  Arms: SGLT2i alone
Drug: Liraglutide or Semaglutide / Dapagliflozin — Combined treatment with Liraglutide 3mg once daily or semaglutide 1mg once weekly subcutaneous injection plus Dapagliflozin 5-10 mg once daily for 6 months.
  Other Names: Combination of GLP1RA and SGLT2i
  Arms: GLP1RA/SGLT2i combination
Drug: Liraglutide or Semaglutide / Dapagliflozin plus intensive weight loss nutrition — Liraglutide 3mg once daily or semaglutide 1mg once weekly subcutaneous injection plus Dapagliflozin 5-10 mg once daily for 6 months combined with intensive lifestyle changes.
  Other Names: Combination of GLP1RA, SGLT2i and intensive weight loss nutrition
  Arms: GLP1RA/SGLT2i combination with intensive lifestyle changes
Other: Usual care — Usual standard care
  Arms: Usual Care

SUMMARY:
As the obesity pandemic continues unabated, one can expect to see an increase in the prevalence of TID/T2D and associated CKD. As a result, death will rise, preceded by an increase in kidney failure, requiring dialysis and renal transplantation. Innovative medical treatment may help prevent chronic kidney disease (CKD) across our healthcare system. The guideline of the American Diabetes Association (ADA) and European Association for the Study of Diabetes (EASD) suggest that patients with obesity, TID/ T2D, and CKD needed either glucagon-like peptide 1 receptor analogs (GLP1-RA) or sodium-glucose cotransport-2 inhibitors (SGLT2i). If neither achieve metabolic control, then the recommendation is to combine both drugs. The evidence base for combining GLP1RA and SGLT2i are not well developed, and hence the impact of the guidelines are limited. This study will provide evidence of discrete metabolic pathways by the GLP1RA/or SGLT2i alone or in combination contributed to metabolic control. The aim of this randomised control trial (RCT) is to test the impact of the combination of GLP1RA/SGLT2i on body weight and kidney damage, in patients with T1DM and CKD. In addition, we will explore associated changes in metabolic pathways with each of the treatments used in the RCT.

DETAILED DESCRIPTION:
Obesity and CKD are linked by obesity-related insulin resistance, a prodromal state associated with impaired glucose tolerance, dyslipidemia, and hypertension, which frequently progresses to overt T1D/T2D. In a seminal 40-year follow-up study in people with a BMI >30kg/m2, the hazard ratio for end-stage kidney disease (ESKD) due to diabetes was 19.4 (95% CI 14.1-26.6). This further supports the role of diabetes in the pathogenesis of CKD. Several complimentary pathological phenomena are postulated to have a mechanistic role in the causal association between obesity, T1D/T2D, and CKD. Excess adiposity precipitate multiple stimuli, including metabolic, hypertensive, and local mechanical stress, which combine to elicit pathogenic responses causing CKD. Changes in volume, structure, and function of adipose tissue contribute to kidney injury through multiple mechanisms. Attendant glucotoxicity can provoke mesangial and tubular cell stress in the kidney through excess glycolysis-driven oxidative stress and the accumulation of advanced glycation end-products. Hyperglycaemia is implicated in the development of glomerular hypertension and hyperfiltration by enhancing proximal tubular sodium reabsorption through sodium-glucose cotransporter-2. This reduces sodium delivery to the macula densa thereby reducing vasoconstrictory tubuloglomerular feedback to the afferent arteriole. Ectopic lipid accumulation in the kidney and the presence of toxic levels of intracellular lipid metabolites (such as ceramide), drive oxidative stress, induce insulin resistance in podocytes, and lead to associated glomerular filtration barrier dysfunction. Adipose tissue stress also causes kidney injury through alterations in the profile of secreted adipokines such as Adiponectin. In humans and rodents, Adiponectin directly supports podocyte health and maintenance of glomerular permselectivity by inducing the expression of the tight junction protein 1 (TJP1) gene (also known as ZO1) and by stimulating fatty acid oxidation and ceramidase activity, which prevents lipotoxicity and oxidative stress. A mechanical role for excess adipose tissue deposition can be posited as a driver of hypertension and kidney injury in obesity. Compression of the kidney parenchyma by expanded perirenal and renal sinus fat lying deep to the renal fascia might promote sodium reclamation by slowing peritubular capillary flow and enhancing tubular solute reabsorption by the counter-current multiplier. This intricate network of metabolic pathways all conspires together to leave many patients with a combination of obesity, T1D/T2D, and CKD. The multitude of these pathways suggests that interventions should simultaneously address as many of these as possible and to date, it is unclear whether GLP1RA/SGLT2i combinations have synergistic benefits pertaining to these pathways.

Many studies have also shown sustained weight loss for decades following bariatric surgery and profound improvements in metabolic control. Weight loss is a dominant mechanism for improving peripheral insulin resistance and glycaemic control after bariatric surgery, but several additional weight-loss-independent mechanisms also contribute.

A meta-analysis of 1913 patients in 7 clinical trials with T2D suggests that GLP1RA/SGLT2i combination therapy had greater reduction in weight of 2.6 kg, HbA1c of 0.6%, and systolic blood pressure of 4.1 mmHg compared to GLP1RA alone and a greater reduction of weight by 1.8 kg, HbA1c by 0.9%, and systolic blood pressure by 2.7 mmHg compared to SGLT2i alone. The studies were not adequately powered to examine CKD or mortality.

Additional analysis of Canagliflozin Cardiovascular Assessment Study (CANVAS) in patients with obesity, T2DM, and CKD used randomized treatment by subgroup interaction to compare the effects of Canagliflozin versus placebo across subgroups defined by baseline use of GLP1RA or not. There were 10,142 patients, of whom 407 (4%) used GLP1RA at baseline. The subgroup of patients with GLP1RA/ SGLT2i combinations had the best outcomes as regards to weight loss, glycaemic improvements, and blood pressure changes compared with the other 3 subgroups (i) no GLP1RA or SGLT2i, (ii) only GLP1RA, and (iii) only SGLT2i. This was the first evidence of a potential synergistic effect of combining GLP1RA and SGLT2i, although there are no trial data specifically designed to describe the effects of this combination. This study together with ADA and EASD guidelines advising clinicians to consider combining GLP1RA and SGLT2i, makes an urgent case for better mechanistic understanding. Identification of such discrete pathways will be a breakthrough.

The aim of this RCT is to test the impact of the combination of GLP1RA/SGLT2i on body weight and kidney damage, in patients with T1DM and CKD. In addition, we will explore associated changes in metabolic pathways with each of the treatments used in the RCT. We will also compare patients in the RCT with patients undergoing bariatric surgery as an exploratory study.

ELIGIBILITY:
Inclusion criteria:

To be considered eligible to participate in this study, a patient must:

* Be aged between 21-65 years,
* Have a BMI ≥ 25 kg/m2,
* Have established diagnosis of Type 1 Diabetes for at least 1 year before screening visit
* Insulin treatment for T1D - may be either via any FDA approved insulin pump (CSII) for at least 6 months prior to screening visit or via multiple daily insulin injections. All participants must be stable on insulin doses/ regimen for at least 3 months
* Have established diagnosis of Chronic Kidney Disease stage 1-4
* Able to give informed consent

Exclusion criteria:

Participants will be excluded if:

* Have been treated with GLP-1 or SGLT2i within the last 3 months and/or have a history of GLP1RA or SGLT2i intolerance
* Diagnosis of T2D or any other type of diabetes (other than type 1)
* Treatment with anti-obesity drugs within 12 weeks prior to randomisation
* Significant changes in the lifestyle (Diet or exercise pattern in within 3 months of the screening visit)
* Any self reported changes (gain or loss) in body weight >5% within 3 months of screening visit
* eGFR ≤15 mL/min/1.73m2
* Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using or willing to use adequate contraceptive methods during the study period
* Experienced diabetic ketoacidosis within 6 months of screening visit
* Experienced sever hypoglycaemia within 6 months of screening visit
* Any of the following laboratory values at screening (liver chemistry > 3X upper limit of normal, high Tg (. 5.7 mmol/L)
* Have terminal illness or are not primarily responsible for their own care
* Any other significant disease or disorder which in the opinion of the investigator, may either put the participants at risk or may influence the result of the study or the participant's ability to participate
* Untreated or uncontrolled hypothyroidism/hyperthyroidism defined as thyroid-stimulating hormone >6 mIU/litre or <0.4 mIU/litre
* Family or personal history of multiple endocrine neoplasia type 2 (MEN2) or familial medullary thyroid carcinoma (FMTC)
* Personal history of non-familial medullary thyroid carcinoma
* History of chronic pancreatitis or idiopathic acute pancreatitis
* Amylase levels three times higher than the upper normal range
* Obesity induced by other endocrinologic disorders (e.g. Cushing's Syndrome)
* Current or history of treatment with medications that may cause significant weight gain, within 12 weeks prior to randomisation, including systemic corticosteroids (except for a short course of treatment, i.e. 7-10 days), atypical antipsychotic and mood stabilizers (e.g. clozapine, olanzapine, valproic acid and its derivatives, and lithium)
* Initiation of antidepressants during the last 12 weeks
* Previous surgical treatment for obesity (excluding liposuction if performed >1 year before trial entry)
* History of other severe psychiatric disorders
* History of known or suspected abuse of alcohol and/or narcotics
* History of major depressive episode during the last 2 years
* Simultaneous participation in other clinical trials of investigational drugs, lifestyle or physical activity interventions. Patients will only be able to take part following participation in a previous clinical trial after a wash-out period of 16 weeks.
* History of dementia or cognitive impairment

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Weight | 26 weeks
  Percentage change in total body weight

SECONDARY OUTCOMES:
Glycaemia | 26 weeks
  Change in HbA1c
Hypertension | 26 weeks
  Change in systolic and diastolic blood pressure
Lipidaemia | 26 weeks
  Change in lipid profile
Albuminuria | 26 weeks
  Change in albumin creatinine ratio
Waist circumference | 26 weeks
  Change in waist circumference
Weight change | 26 weeks
  Proportion of participants reaching total body weight loss of ≥5%, ≥10% and ≥15%

CONTACTS AND LOCATIONS:
Overall Officials: Ebaa Al Ozairi, Principal Investigator — Dasman Institute
Locations (1):
- Dasman Diabetes Institute, Kuwait City, Al Asimah, Kuwait

REFERENCES:
- [Derived] Al-Ozairi E, Narula K, Miras AD, Taghadom E, Samad AE, Al Kandari J, Alyosef A, Mashankar A, Al-Najim W, le Roux CW. Obesity Treatments to Improve Type 1 Diabetes (OTID): a randomized controlled trial of the combination of glucagon-like peptide 1 analogues and sodium-glucose cotransporter 2 inhibitors-protocol for Obesity Treatments to Improve Type 1 Diabetes (the OTID trial). Trials. 2024 Feb 16;25(1):129. doi: 10.1186/s13063-024-07930-3. PMID 38365744

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-12-11): https://cdn.clinicaltrials.gov/large-docs/07/NCT05390307/SAP_000.pdf